CLINICAL TRIAL: NCT06066086
Title: A Hinge Flap as an Additional Layer to Reinforce the Buccal Advancement Flap for Treating Chronic Oroantral Fistulae (COAF) in the Most Posterior Aspect of the Maxilla"
Brief Title: A Hinge Flap to Reinforce Buccal Advancement Flap
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Ghada Amin Khalifa, PhD, Professor of Oral and Maxillofacial Surgery, Qassim University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID: 23-24-14
Record Dates: First submitted 2023-04-24; First posted 2023-10-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-09

CONDITIONS: Oroantral Fistula
Keywords: Chronic Oroantral Fistula
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hinge Flap group (Experimental): Patients who will be included in this study will be treated by using hinge flap and buccal advancement flap to close their oroantral fistula. A circular incision will be performed at the oral side of the oroantral fistula. The tissues will be reflected and sutured by purse sutures. Then the tissues will be pushed up to close sinus membrane. A pyramidal flap will be reflected at the buccal tissues, then horizontal incisions will be performed at the base of the flap to allow advancement of the flap over the fistula and a tension-free suturing to the palatal tissues.
  Interventions: Procedure: A hinge flap will be performed to reinforce the buccal advancement flap to close the oroantral fistula at the most posterior area of the maxilla
- Palatal Flap group (Active Comparator): Patients who will be included in this study will be treated by using he anteriorly based palatal rotational flap to close the oroantral fistula. Two paralleling incisions will be performed on the palatal side of the fistula. The distance between the two incisions will be 2 to 3 mm greater than the width of the fistula. Then the two incisions will be connected together via a circular incision at the bony end of the hard palate. The flap reflection will be performed, and the greater palatine vessels will be legated and cauterized to allow lateral repositioning of the flap over the fistula. The flap will be sutured to the buccal tissues.
  Interventions: Procedure: An anteriorly based palatal flap will be performed to close the oroantral fistula at the most posterior area of the maxilla

INTERVENTIONS:
Procedure: A hinge flap will be performed to reinforce the buccal advancement flap to close the oroantral fistula at the most posterior area of the maxilla — The hinge flap is raised via circular incision around the oral side of the oroantral fistula then sutured with purse suture to close the sinus membrane perforation and it is used as an additional layer that reinforce the buccal advancement flap
  Arms: Hinge Flap group
Procedure: An anteriorly based palatal flap will be performed to close the oroantral fistula at the most posterior area of the maxilla — Two paralleling incisions will be performed on the palatal side of the fistula. The distance between the two incisions will be 2 to 3 mm greater than the width of the fistula. Then the two incisions will be connected together via a circular incision at the bony end of the hard palate. The flap reflection will be performed, and the greater palatine vessels will be legated and cauterized to allow lateral repositioning of the flap over the fistula. The flap will be sutured to the buccal tissues.
  Arms: Palatal Flap group

SUMMARY:
Background The chronic oroantral fistulas (COAF) is an epithelized communication that is formed between the squamous epithelium of the oral cavity and the pseudo-stratified columnar ciliated epithelium of the maxillary sinus with a high recurrent rate. The use of palatal flaps has been documented for treating such fistulae. The presence of the oroantral fistula at the area of second molars or maxillary tuberosity could complicate the use of the palatal rotational flap where the arch of its rotation is increased leading to compromised blood supply. The use of the buccal flap is not advocated because it is very thin.

Rationale Double or triple-layer closure is indicated to avoid recurrence of the COAF. Different layers have been documented to minimize the risk of recurrence and reinforce buccal flaps. The oral tissues at the oral side of the oroantral fistula could used as an additional layer with buccal advancement flap and buccal fat to omit the use of palatal flap with its subsequent problems in the most posterior aspect of the maxilla Study objectives Therefore, this study will be conducted to evaluate the use of hinge flaps to reinforce the buccal advancement flap for surgical closure of the COAF in the most posterior area of the maxilla

Methods The hinge flap will be performed at the oral side of the COAF to close the perforation in the sinus membrane. The oral side of the COAF will be closed with buccal advancement flap. The success rate, recurrence, time of surgery, postoperative complications, will be evaluated.

DETAILED DESCRIPTION:
Background:

The surgical therapy of COAF is one of the most challenging subjects. Local flaps are usually performed to close oroantral fistula (OAF). Each flap has advantages and limitations; none is superior to others. The appropriate flap is determined by the location and size of OAF, prosthetic therapy, and the surgeon's skill.5 Buccal advancement flaps, palatal rotational flaps, and buccal fat pad (BFP) are the most commonly employed local flaps, either alone or in combination. Although buccal flap surgery is easy, it is not recommended for large, COAFs because it is very thin, has poor perfusion, and is prone to strain due to lip and check muscle movements, making it more prone to rupture and tear.The palatal rotational flap is preferred in such instances, however, it has significant technical challenges, such as bunching the flap along its axis of rotation and kinking the greater palatine artery. If the OAFs are in the most posterior area of the maxilla, particularly towards the second and third molars, flap rotation may jeopardize the vascular pedicle, resulting in closure failure. So, many authors supported the use of BFP to add strength to the buccal flap, but it also has significant drawbacks.6 First, the BFP can be perforated and detached from its blood supply while being dissected from its surrounding components, resulting in necrosis. Furthermore, in certain instances, the size of the BFP may be insufficient to cover the OAF.

Rationale A prospective study will be enrolled to evaluate the use of the hinge flap to reinforce the buccal advancement flap for the management of COAFs in the most posterior area of the maxilla. The second aim of the study was to implement an algorithm for the management of OAFs based on the authors' 20 years of experience in the management of OAFs.

Methods A double-blinded randomized control trial will be conducted. Patients were divided into two groups: hinge flap or palatal flap. The palatal flap group will be served as the control group, while the hinge flap will be the tested group.The patient sequences will be used for randomization. Patients with even numbers will be assigned to the hinge flap group, while those with odd numbers will be assigned to the palatal flap group. The following steps will be taken to achieve blindness: 1) The patients and evaluators who will interview them to measure the study's variables will not informed about the study and 2) The investigators who will review the questionnaires and the statistician who will analyze the study's results will know the study's groups as A and B.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic oroantral fistula at the most posterior area of the maxilla
2. Ages above 18 years
3. Patients who are medical free

Exclusion Criteria:

1. Oroantral communications
2. Absence of sinus infection
3. Oroantral fistula which are resulted from tumor resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of Surgery | 30 minutes
  The time elapsed from the initial incision to final closure of the flap. The time will be calculated in minutes. The mean and standard deviation will be then calculated and used to compare between the study's arms.A prolonged time means worse outcomes
Difficulties during surgeries | 60 minutes
  Surgical difficulties scoring system will be used.Surgical difficulty was assessed by the operator using an index of 1-10 with the following divisions: 1-3 low difficulty, 4-6 intermediate difficulty, and 7-10 high difficulty. A low difficulty score means a better outcome
Recurrence of the Oroantral fistula | At the end of the postoperative fourth month
  The patients will be followed after surgery for the success or failure of the surgical closure. The follow-up will be weekly in the first month, and then monthly in the next three months.The recurrence means worse outcomes

SECONDARY OUTCOMES:
Patients' satisfaction | At the end of the fourth month after surgery
  A patient satisfaction survey is a set of questions used to collect feedback from patients to measure their satisfaction with the quality and care of the healthcare service provider.Based on their responses, patients will be divided into three categories: Promoters (9-10), Passives (7-8), and Detractors (0-6).

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A khalifa, Professor, Study Director — Department of Maxillofacial Study and Diagnostic Sciences, College of Dentistry, Qassim University
Locations (1):
- College of Dentistry, Qassim University, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No